CLINICAL TRIAL: NCT03290248
Title: A Prospective, Controlled, Double Blind, Multi-Center, Randomized, 3 Arm, Phase 1b/2a Study to Assess the Safety, Tolerability, and Preliminary Efficacy of B244 Delivered as an Intranasal Spray in Healthy Volunteers and Subjects With Seasonal Allergic Rhinitis
Brief Title: Study to Assess the Safety, Tolerability, and Preliminary Efficacy of B244 in Healthy Volunteers and Subjects With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: Orange County Research Center (Other); Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARB244-001
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis; Allergic Rhinitis Due to Grass Pollen; Healthy Volunteers
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1:1 so that equal number of subjects will be treated in each arm of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Interventions: Biological: Vehicle
- B 244 1x (low dose) (Active Comparator): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Interventions: Biological: B244 suspension
- B244 4x (mid dose) (Active Comparator): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Interventions: Biological: B244 suspension

INTERVENTIONS:
Biological: B244 suspension — B244 suspension in 30ml/bottle
  Arms: B 244 1x (low dose); B244 4x (mid dose)
Biological: Vehicle — Vehicle, 30ml/bottle
  Arms: Vehicle

SUMMARY:
This is a Prospective, Controlled, Double Blinded, Single Center, Randomized, 3 Arm, Parallel Assignment, Phase 1b/2a Study to assess the safety, tolerability, and preliminary efficacy of B244 delivered as an intranasal spray in healthy volunteers and subjects with seasonal allergic rhinitis.

DETAILED DESCRIPTION:
This is a Prospective, Controlled, Double Blinded, Single Center, Randomized, 3 Arm, Parallel Assignment, Phase 1b/2a Study to assess the safety, tolerability, and preliminary efficacy of B244 delivered as an intranasal spray in healthy volunteers and subjects with seasonal allergic rhinitis. This will be a 2-part study. In Part 1, safety and tolerability will be evaluated during 14 days of study treatment twice-a-day followed by 4 weeks of follow-up in healthy volunteers. In Part 2, preliminary efficacy will be evaluated in subjects with a history of seasonal allergic rhinitis outside of the local pollen season.

For Part 1 (safety and tolerability evaluation in healthy volunteers) we will enroll 24 subjects. Safety and tolerability will be assessed by reporting of AEs, physical examination and vital signs (blood pressure, heart rate, respiratory rate) during 14 days of treatment and up to 28 days of follow-up.

An internal safety committee meeting will review the 2 week Part 1 safety data and, if there are no safety concerns, the study will proceed to Part 2 to evaluate preliminary efficacy in subjects with a history of seasonal allergic rhinitis (SAR)

For Part 2 (preliminary efficacy evaluation in subjects with a history of SAR to ragweed pollen) will enroll 42 subjects. Safety and tolerability will be assessed in subjects with allergic rhinitis by reporting of AEs, physical examination and vital signs (blood pressure, heart rate, respiratory rate) during 14 days of treatment.

For Part 2, study will be paused for safety review using the same stopping criteria as in Part 1.

Rescue medications will not be allowed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 18 to 65 years of age (committed to consistent use of an acceptable method of birth control as described in Section 10).
* In good general health as determined by a thorough medical history and physical examination, and vital signs.
* Nonsmoker or ex-smoker (stopped >1 year prior to study entry).
* Subjects willing and able to provide written informed consent.
* Is willing and able to comply with the requirements of the protocol and must be available for the full duration of the study.
* For Part 1, subjects asymptomatic from any seasonal or perennial allergens.
* For Part 1, elevated systolic blood pressure greater than 120 but less than 160 and never been on antihypertensive medications or have been off any hypertensive treatment for a period of 12 weeks or longer.
* For Part 2, subjects with a well-documented history of seasonal allergic rhinitis (specifically ragweed pollen) with documentation of sensitivity by positive skin testing and/or IgE testing to the relevant allergens 12 months prior to enrollment that correlate with clinical history.
* For Part 2, a ragweed positive skin prick test with a wheal diameter at least 5 mm larger than the negative control and/or a ragweed specific IgE greater or equal to 0.7 kU/L.
* For Part 2, subjects with confounding allergies, or sensitization to cat epithelia, dog epithelia, Dermatophagoides farinae, or Dermatophagoides pteronyssinus or prevalent and relevant seasonal allergens as per the skin prick test may be included if sensitization is not clinically relevant (ie. subject is non-symptomatic and/or can avoid the allergen during the study) at the discretion of the Investigator.
* For Part 2, subjects with a baseline TNSS ≤ 3/12 at Visit 3 and a minimum qualifying TNSS score of a change of 6/12 from their baseline score after NAC #1 on at least 2 diary cards.
* For Part 2, subjects' average post diluents nasal congestion score must be < 1 at admission for each study visit.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Female of childbearing potential not using adequate contraceptive measures.
* Smoking within the past year or during the protocol.
* Systemic corticosteroid or other immunosuppressive medications use in the previous three months or during the protocol.*
* Intranasal corticosteroid use in the previous month or during the protocol.*
* Intranasal antihistamine or cromolyn use in the previous week or during the study.*
* Allergen immunotherapy during previous 12 months or during the protocol.*
* Omalizumab use in previous 12 months or during the protocol.*
* Systemic antihistamine or leukotriene modifying medication use in the previous week or during the protocol.*
* Use of antibiotics, NSAIDS, antihypertensives, beta-blockers, photosensitizing medications, or vitamin D supplements during study.
* Use of any intranasally administered over-the-counter product or nasal irrigation (e.g., neti pot) during study.
* Inability to give informed consent.
* Persistent asthma or any medical condition that in the opinion of the investigator may compromise the subject's ability to safely participate in the study.
* Subjects with any significant clinical abnormalities which may interfere with study participation.
* Prior use of AO+ Mist.
* Subjects with immunodeficiencies, nasal lesions, nasal polyps, or sinus infections.
* Use of an investigational drug within 30 days before screening Visit 1. * Exclusionary criterion due to 1) medication use as marker of persistent comorbid allergic or inflammatory condition that may increase subject risk with study participation, 2) potential of medication to interfere with study outcome measures or results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Study PI
Locations (2):
- Orange County Research Center, Tustin, California, United States
- Inflamax, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle: Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Vehicle: Vehicle, 30ml/bottle
- B 244 1x (Low Dose): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (1x10E9 cells/ml) in 30ml/bottle
- B244 4x (Mid Dose): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
Period: Study Part 1
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Study Part 2
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Started | 15 | 16 | 16
Completed | 15 | 16 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population includes patients from Part 1 (n=24) Part 2 (n=47) of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose) | Total
Number analyzed (Participants) | 23 | 24 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  years
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1 | 47.29 (11.179) | 44.60 (11.193) | 45.36 (10.316) | 45.76 (10.477)
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2 | 47.20 (9.470) | 45.49 (12.145) | 42.30 (12.754) | 44.95 (11.516)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  Participants
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1: Female | 3 | 5 | 3 | 11
    Part 1: Male | 5 | 3 | 5 | 13
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2: Female | 10 | 12 | 9 | 31
    Part 2: Male | 5 | 4 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  Participants
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1: Hispanic or Latino | 3 | 5 | 5 | 13
    Part 1: Not Hispanic or Latino | 5 | 2 | 1 | 8
    Part 1: Unknown or Not Reported | 0 | 1 | 2 | 3
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2: Hispanic or Latino | 3 | 1 | 3 | 7
    Part 2: Not Hispanic or Latino | 12 | 15 | 13 | 40
    Part 2: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  Participants
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Part 1: Asian | 0 | 1 | 2 | 3
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Part 1: Black or African American | 2 | 2 | 1 | 5
    Part 1: White | 6 | 5 | 5 | 16
    Part 1: More than one race | 0 | 0 | 0 | 0
    Part 1: Unknown or Not Reported | 0 | 0 | 0 | 0
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2: American Indian or Alaska Native | 1 | 0 | 0 | 1
    Part 2: Asian | 3 | 2 | 6 | 11
    Part 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Part 2: Black or African American | 5 | 9 | 5 | 19
    Part 2: White | 6 | 5 | 5 | 16
    Part 2: More than one race | 0 | 0 | 0 | 0
    Part 2: Unknown or Not Reported | 0 | 0 | 0 | 0
Tobacco History [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  Participants
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1: Never | 8 | 8 | 5 | 21
    Part 1: Current | 0 | 0 | 0 | 0
    Part 1: Former | 0 | 0 | 3 | 3
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2: Never | 12 | 16 | 16 | 44
    Part 2: Current | 0 | 0 | 0 | 0
    Part 2: Former | 3 | 0 | 0 | 3
Screening Height [Mean (Standard Deviation); unit: cm] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  cm
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1 | 174.0 (8.20) | 169.8 (8.40) | 172.8 (11.60) | 172.2 (9.24)
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2 | 169.0 (3.73) | 165.9 (8.38) | 167.1 (9.88) | 167.3 (8.39)
Screening Weight [Mean (Standard Deviation); unit: kg] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  kg
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1 | 81.83 (22.316) | 77.94 (10.679) | 89.55 (21.376) | 83.10 (18.699)
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2 | 76.89 (15.279) | 79.69 (14.577) | 79.72 (17.633) | 78.81 (15.604)
Screening BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Part 1 and Part 2 were of different patient populations. Baseline demographic metrics were collected separately for each part.
  kg/m^2
    Part 1: number analyzed (Participants) | 8 | 8 | 8 | 24
    Part 1 | 26.77 (5.890) | 27.15 (4.197) | 29.76 (5.013) | 27.89 (5.046)
    Part 2: number analyzed (Participants) | 15 | 16 | 16 | 47
    Part 2 | 26.86 (4.803) | 28.93 (4.868) | 28.59 (6.053) | 28.15 (5.250)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all treatment-related adverse events reporting during the study duration for subjects only from Part 1 of the study.
Time Frame: Baseline to Day 28
Population: Population included subjects from Part 1 of the study and those who had received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Drug Related TEAE | 0 | 0 | 0
  Drug Related Severe TEAE | 0 | 0 | 0
  Drug Related Serious TEAE | 0 | 0 | 0

2. Secondary Outcome: Change in Total Nasal Symptom Score (TNSS) After Prophylaxis Treatment
Description: Total Nasal Symptom Score (TNSS) is the sum of sub-scores for each of nasal congestion, sneezing, nasal itching, and rhinorrhea at each time point, using a four point scale (0-3; 0 = none; 1 = mild; 2 = moderate; 3 = severe), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the sub-score for each of the symptoms to a total out of 12. For TNSS and Area Under the Curve (AUC) analyses, an Analysis of Covariance with treatment and site as factors and Visit 3 (or Visit 2) value as a covariate was used to test for treatment effect at Visit 4.
  Observed AUC (0-2 Hours) was defined as TNSS from 0 to 120 minutes post Nasal Allergen Challenge (NAC). The Pre-NAC Adjusted AUC (0-2 Hours) was defined as the observed value minus the 0 minutes prior NAC value.
Time Frame: Visit 3 (or alternative baseline at Visit 2) to Visit 4 (14 days prophylaxis treatment). Visit 2 was used as an alternate baseline to report baseline values prior to any nasal allergen challenge (NAC) to minimize any potential priming effects.
Population: Population includes only patients from Part 2 of the study.
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
score on a scale*hours
  Observed AUC (0-2 Hours) | -5.1 (3.53) | -2.5 (4.51) | -4.9 (3.66)
  Pre-NAC Adjusted (0-2 Hours) | -5.9 (3.88) | -3.7 (6.84) | -4.9 (3.29)

3. Secondary Outcome: Subjective Nasal Symptom Scores of Nasal Congestion After Prophylaxis Treatment
Description: All measurements were taken 120 minutes Post-Nasal Allergen Challenge (Post-NAC) at Visit 4 and compared to Baseline Visit 3. Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline. Nasal congestion was categorized as None, Mild, Moderate, or Severe.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Visit 2 (Day 0): None | 4 | 2 | 5
  Visit 2 (Day 0): Mild | 8 | 6 | 4
  Visit 2 (Day 0): Moderate | 0 | 5 | 4
  Visit 2 (Day 0): Severe | 3 | 3 | 3
  Visit 3 (Day 14): None | 3 | 4 | 4
  Visit 3 (Day 14): Mild | 4 | 3 | 4
  Visit 3 (Day 14): Moderate | 6 | 5 | 5
  Visit 3 (Day 14): Severe | 2 | 4 | 3
  Visit 4 (Day 28): None | 3 | 4 | 7
  Visit 4 (Day 28): Mild | 8 | 6 | 6
  Visit 4 (Day 28): Moderate | 3 | 3 | 3
  Visit 4 (Day 28): Severe | 1 | 3 | 0

4. Secondary Outcome: Subjective Nasal Symptom Scores of Rhinorrhea After Prophylaxis Treatment
Description: All measurements were taken 120 minutes Post-Nasal Allergen Challenge (Post-NAC) at Visit 4 and compared to Baseline Visit 3. Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline. Rhinorrhea was categorized as None, Mild, Moderate, or Severe.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Groups:
- B244 4x (Mid Dose): Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (4x10E9 cells/ml)in 30ml/bottle
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Visit 2 (Day 0): None | 8 | 9 | 8
  Visit 2 (Day 0): Mild | 2 | 5 | 4
  Visit 2 (Day 0): Moderate | 3 | 0 | 3
  Visit 2 (Day 0): Severe | 2 | 2 | 1
  Visit 3 (Day 14): None | 5 | 6 | 6
  Visit 3 (Day 14): Mild | 6 | 5 | 5
  Visit 3 (Day 14): Moderate | 3 | 1 | 3
  Visit 3 (Day 14): Severe | 1 | 4 | 2
  Visit 4 (Day 28): None | 11 | 10 | 10
  Visit 4 (Day 28): Mild | 2 | 3 | 4
  Visit 4 (Day 28): Moderate | 2 | 1 | 2
  Visit 4 (Day 28): Severe | 0 | 2 | 0

5. Secondary Outcome: Subjective Nasal Symptom Scores of Nasal Itching After Prophylaxis Treatment
Description: All measurements were taken 120 minutes Post-Nasal Allergen Challenge (Post-NAC) at Visit 4 and compared to Baseline Visit 3. Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline. Nasal itching was categorized as None, Mild, Moderate, or Severe.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Visit 2 (Day 0): None | 6 | 10 | 10
  Visit 2 (Day 0): Mild | 4 | 4 | 2
  Visit 2 (Day 0): Moderate | 2 | 1 | 3
  Visit 2 (Day 0): Severe | 3 | 1 | 1
  Visit 3 (Day 14): None | 6 | 7 | 9
  Visit 3 (Day 14): Mild | 4 | 5 | 4
  Visit 3 (Day 14): Moderate | 5 | 3 | 2
  Visit 3 (Day 14): Severe | 0 | 1 | 1
  Visit 4 (Day 28): None | 11 | 11 | 13
  Visit 4 (Day 28): Mild | 4 | 3 | 3
  Visit 4 (Day 28): Moderate | 0 | 1 | 0
  Visit 4 (Day 28): Severe | 0 | 1 | 0

6. Secondary Outcome: Subjective Nasal Symptom Scores of Sneezing After Prophylaxis Treatment
Description: All measurements were taken 120 minutes Post-Nasal Allergen Challenge (Post-NAC) at Visit 4 and compared to Baseline Visit 3. Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline. Sneezing was categorized as None, Mild, Moderate, or Severe.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Visit 2 (Day 0): None | 9 | 13 | 11
  Visit 2 (Day 0): Mild | 5 | 3 | 3
  Visit 2 (Day 0): Moderate | 1 | 0 | 2
  Visit 2 (Day 0): Severe | 0 | 0 | 0
  Visit 3 (Day 14): None | 9 | 13 | 13
  Visit 3 (Day 14): Mild | 5 | 1 | 1
  Visit 3 (Day 14): Moderate | 1 | 2 | 1
  Visit 3 (Day 14): Severe | 0 | 0 | 1
  Visit 4 (Day 28): None | 10 | 13 | 13
  Visit 4 (Day 28): Mild | 5 | 3 | 3
  Visit 4 (Day 28): Moderate | 0 | 0 | 0
  Visit 4 (Day 28): Severe | 0 | 0 | 0

7. Secondary Outcome: Nasal Symptom-free Response Rate in Nasal Congestion Scores After Prophylaxis Treatment
Description: Nasal symptom free response rate was assessed 120 minutes Post-Nasal Allergen Challenge (Post-NAC) to be scored as Yes or No to nasal congestion at Visit 4 (yes indicates subject is free from nasal congestion symptom and no indicates subject still has nasal itching symptom). Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Yes | 3 | 4 | 7
  No | 12 | 12 | 9

8. Secondary Outcome: Nasal Symptom-free Response Rate in Rhinorrhea Scores After Prophylaxis Treatment
Description: Nasal symptom free response rate was assessed 120 minutes Post-Nasal Allergen Challenge (Post-NAC) to be scored as Yes or No to rhinorrhea at Visit 4 (yes indicates subject is free from rhinorrhea symptom and no indicates subject still has nasal itching symptom). Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Yes | 11 | 10 | 10
  No | 4 | 6 | 6

9. Secondary Outcome: Nasal Symptom-free Response Rate in Nasal Itching Scores After Prophylaxis Treatment
Description: Nasal symptom free response rate was assessed 120 minutes Post-Nasal Allergen Challenge (Post-NAC) to be scored as Yes or No to nasal itching at Visit 4 (yes indicates subject is free from nasal itching symptom and no indicates subject still has nasal itching symptom). Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Yes | 11 | 11 | 13
  No | 4 | 5 | 3

10. Secondary Outcome: Nasal Symptom-free Response Rate in Sneezing Scores After Prophylaxis Treatment
Description: Nasal symptom free response rate was assessed 120 minutes Post-Nasal Allergen Challenge (Post-NAC) to be scored as Yes or No to sneezing at Visit 4 (yes indicates subject is free from sneezing symptom and no indicates subject still has nasal itching symptom). Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Yes | 10 | 13 | 13
  No | 5 | 3 | 3

11. Secondary Outcome: Nasal Symptom-free Response Rate in TNSS After Prophylaxis Treatment
Description: Number of subjects that had 25% and 50% reduction in Observed Area Under the Curve (AUC) (0-120 minutes)/Pre-NAC Adjusted AUC (0-120 minutes) at Visit 4 (Day 28) from Visit 2 Observed AUC (0-120 minutes)/Pre-NAC Adjusted AUC (0-120 minutes). For TNSS and Area Under the Curve (AUC) analyses, an Analysis of Covariance with treatment and site as factors and Visit 3 (or Visit 2) value as a covariate was used to test for treatment effect at Visit 4. Observed AUC (0-2 Hours) was defined as TNSS from 0 to 120 minutes post Nasal Allergen Challenge (NAC). The Pre-NAC Adjusted AUC (0-2 Hours) was defined as the observed value minus the 0 minutes prior NAC value.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  25% Reduction from Visit 2 Observed AUC (0-120 minutes): Yes | 9 | 6 | 12
  25% Reduction from Visit 2 Observed AUC (0-120 minutes): No | 6 | 10 | 4
  25% Reduction from Visit 2 Pre-NAC Adjusted AUC (0-120 minutes): Yes | 9 | 8 | 15
  25% Reduction from Visit 2 Pre-NAC Adjusted AUC (0-120 minutes): No | 6 | 8 | 1
  50% Reduction from Visit 2 Observed AUC (0-120 minutes): Yes | 3 | 3 | 6
  50% Reduction from Visit 2 Observed AUC (0-120 minutes): No | 12 | 13 | 10
  50% Reduction from Visit 2 Pre-NAC Adjusted AUC (0-120 minutes): Yes | 7 | 6 | 8
  50% Reduction from Visit 2 Pre-NAC Adjusted AUC (0-120 minutes): No | 8 | 10 | 8

12. Other Pre Specified Outcome: Change in Peak Nasal Inspiratory Flow (PNIF)
Description: Peak Nasal Inspiratory Flow (PNIF) is a commonly used method for assessing nasal patency and provides an objective measurement of nasal airflow obstruction. The outcome is a direct representation of nasal congestion. Change in PNIF Observed Inverted Area Under the Curve (AUC) was measured between baseline and Visit 4. A decrease in PNIF Observed Inverted AUC(0-2 Hours) was considered an improvement in nasal airflow obstruction. Visit 3 was considered Baseline. Visit 2 was considered an alternate Baseline.
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Mean (Standard Deviation); unit: L*Hr/min
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
L*Hr/min
  Change from Visit 3 to Visit 4 | -60.8 (57.83) | -8.6 (39.62) | -60.9 (57.48)
  Change from Visit 2 to Visit 4 | -51.2 (99.99) | -30.4 (96.76) | -59.8 (57.77)

13. Other Pre Specified Outcome: Nasal Inflammation Score Using Otoscope
Description: Nasal inflammation were graded by a clinician using a 0-3 nasal inflammation scale based on otoscope measurement where 0 = none, 1 = mild, 2 = moderate, and 3 = severe inflammation 120 minutes Post Nasal Allergen Challenge (Post-NAC).
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Visit 3 (Day 14): None | 0 | 0 | 0
  Visit 3 (Day 14): Mild | 5 | 4 | 8
  Visit 3 (Day 14): Moderate | 8 | 10 | 8
  Visit 3 (Day 14): Severe | 2 | 2 | 0
  Visit 4 (Day 28): None | 2 | 2 | 6
  Visit 4 (Day 28): Mild | 9 | 9 | 5
  Visit 4 (Day 28): Moderate | 3 | 4 | 5
  Visit 4 (Day 28): Severe | 1 | 1 | 0

14. Other Pre Specified Outcome: Intranasal Nitric Oxide Levels
Description: Exhaled nasal nitric oxide (NO) was measured from the nasal cavity by a NO analyzer 120 minutes Post Nasal Allergen Challenge (Post-NAC).
Time Frame: as for outcome 2
Population: Population includes only patients from Part 2 of the study.
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 7 | 8 | 8
ppb
  Visit 3 (Day 14) | 61.9 (57.77) | 33.9 (26.68) | 81.9 (104.88)
  Visit 4 (Day 28) | 63.6 (55.42) | 27.3 (25.25) | 52.7 (41.13)

15. Other Pre Specified Outcome: Change in Cytokine Concentration in Nasal Cavity and Blood
Description: To evaluate if B244 administration will affect the levels of cytokine biomarkers in nasal cavity and blood.
Time Frame: as for outcome 2
Population: Data was not collected for this exploratory endpoint.
Arm/Group | Vehicle | B 244 1x (Low Dose) | B244 4x (Mid Dose)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: Baseline to end of study (Day 42). Part 2: Baseline to end of study (Day 28).
Description: Population included subjects from Part 1 (n=24) and Part 2 (n=47) of the study and those who received at least 1 dose of IP. All clinical events were to be recorded in the CRF. AEs resulting from concurrent illnesses or reactions to concurrent medications were also to be recorded. Each adverse clinical event was evaluated for duration, intensity, and whether the event may be associated with the IP or other causes. AEs believed to be possibly related to IP must be followed until resolution.
Groups:
- Part 1: Vehicle: Part 1
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Vehicle: Vehicle, 30ml/bottle
- Part 1: B244 1x (Low Dose): Part 1
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (1x10E9 cells/ml) in 30ml/bottle
- Part 1: B244 4x (Mid Dose): Part 1
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
- Part 2: Vehicle: Part 2
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  Vehicle: Vehicle, 30ml/bottle
- Part 2: B244 1x (Low Dose): Part 2
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (1x10E9 cells/ml) in 30ml/bottle
- Part 2: B244 4x (Mid Dose): Part 2
  Intranasal application:
  1 pump (140ul) per nostril BID for 14 days
  B244 suspension: B244 suspension (4x10E9 cells/ml) in 30ml/bottle
Arm/Group | Part 1: Vehicle | Part 1: B244 1x (Low Dose) | Part 1: B244 4x (Mid Dose) | Part 2: Vehicle | Part 2: B244 1x (Low Dose) | Part 2: B244 4x (Mid Dose)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 1/8 | 1/15 | 0/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Vehicle (N=8) | Part 1: B244 1x (Low Dose) (N=8) | Part 1: B244 4x (Mid Dose) (N=8) | Part 2: Vehicle (N=15) | Part 2: B244 1x (Low Dose) (N=16) | Part 2: B244 4x (Mid Dose) (N=16)
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish or otherwise publicly disclose the analyzed study data and conclusions drawn from the study.

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT03290248/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT03290248/SAP_001.pdf